CLINICAL TRIAL: NCT00847639
Title: Evaluation of Lenalidomide as Maintenance Therapy Post Allogeneic Hematopoietic Cell Transplantation for High-risk Multiple Myeloma
Brief Title: Safety Study of Lenalidomide Maintenance Therapy Post Allogeneic HCT for High-risk Multiple Myeloma
Acronym: 07-REV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-REV
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; lenalidomide; Revlimid; Allogeneic Hematopoietic Cell Transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide maintenance therapy will start within 60 to 180 days after allogeneic HCT at a starting dose of 10mg PO once daily. Dose escalation and de-escalation are performed depending on tolerability of lenalidomide. The dose range is 5mg every other day and 5 to 25 mg daily from days 1-21 followed by 7 days of rest for 12 cycles (each cycle 28 days).
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — Lenalidomide maintenance therapy will start within 60 to 90 days after allogeneic HCT at a starting dose of 10mg PO once daily.
  Dose escalation and de-escalation are performed depending on tolerability of lenalidomide.
  The dose range is 5mg every other day and 5 to 25 mg daily from days 1-21 followed by 7 days of rest for 12 cycles (each cycle 28 days).
  Other Names: Revlimid

SUMMARY:
This is a multi-institution, non-randomized, open label, Phase IIa prospective trial to evaluate the safety and tolerability of maintenance lenalidomide after allogeneic hematopoietic stem cell transplantation (HCT).

Lenalidomide maintenance therapy will start between day 60 and 90 after allogeneic HCT at a starting dose of 10mg PO once daily. Dose escalation and de-escalation will be performed depending on tolerability of lenalidomide. Dose range is 5mg every other day to 5 - 25 mg given daily on days 1-21 of a 28-day cycle for 12 cycles maximum or maximum of 12 months from first dose of study drug.

Patients will be followed until 28 days from completing the 12th planned cycle of lenalidomide maintenance or 12 months from first dose of study drug, which ever comes first, (14 to 15 months after receiving the allograft) or discontinuation of study drug.

ELIGIBILITY:
Inclusion Criteria:

* One prior allograft from an 8/8 or 7/8 allele matched related or unrelated donor, received 60 to 90 days prior to initiation of lenalidomide
* Meet the diagnostic criteria of symptomatic myeloma at anytime prior to allogeneic HCT
* Have high-risk multiple myeloma
* Received ≤ three (3) prior lines of therapy. Prior therapies may include: combination chemotherapy, monotherapy, lenalidomide and autologous HCT. Localized radiation therapy does not count as a single line of therapy. Previous progression on lenalidomide does not exclude participation in the study.
* Received a reduced intensity conditioning regimen
* Received or are receiving a GVHD prophylaxis regimen of a calcineurin inhibitor in combination with either methotrexate, mycophenolate mofetil (MMF) or sirolimus
* Karnofsky performance score ≥ 80 or ECOG ≤ 2
* There must be at least 50% donor chimerism and no evidence of falling donor chimerism within 1 month of enrollment
* Laboratory test results within range, within 14 days prior to initiation of lenalidomide
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.

Exclusion Criteria:

* Disease progression at time of study entry
* Patients with any grade III-IV GVHD at the time of study entry
* Patients requiring additional immunosuppressive therapy to control acute GVHD other than corticosteroids and immunosuppressive agents used for prophylaxis.
* Concomitant use of other investigational agents
* Patients who have received donor lymphocyte infusions
* Active CNS malignancy
* Uncontrolled bacterial, viral, or fungal infections
* Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ < 5 years from study entry.
* Known hypersensitivity or desquamating rash to either thalidomide or lenalidomide.
* Known positive for HIV or active infectious hepatitis.
* Women who are pregnant or breastfeeding.
* New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2013-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To determine tolerability and safety profile of a maximum of 12 cycles or 12 months from first dose (which ever comes first) of lenalidomide maintenance therapy post allogeneic hematopoietic cell transplantation for high risk multiple myeloma. | 12 months

SECONDARY OUTCOMES:
To estimate the incidences of ≥ grade 3 adverse events, graft failure, infections, treatment-related mortality (TRM) and incidence and severity of acute and chronic GVHD after initiation of lenalidomide. | 13 months
To measure the overall response and best response rates to lenalidomide maintenance therapy following allogeneic HCT. | 13 Months
To determine time to disease progression and overall survival after lenalidomide. | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Alsina, MD, Principal Investigator — H. Lee Moffitt Cancer Center; Marcelo Pasquini, MD, Study Chair — CIBMTR/ Medical College of Wisconsin
Locations (8):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Pennsylvania Hospital Center, Philadelphia, Pennsylvania
  - The University of Texas, M.D. Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin